CLINICAL TRIAL: NCT05663658
Title: External Oblique Intercostal Plane Block for Postoperative Analgesia in Obese Patients Undergoing Laparoscopic Sleeve Gastrectomy
Brief Title: External Oblique Intercostal Plane Block for Laparoscopic Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: anestezi1
Record Dates: First submitted 2022-12-15; First posted 2022-12-23 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-01

CONDITIONS: Obesity; Analgesia; Postoperative Pain
MeSH Terms: conditions — Obesity; Agnosia; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): The patients in Control Group will be received patient controlled analgesia with morphine for postoperative analgesia
  Interventions: Other: Intravenous morphine patient control device
- External oblique intercostal plane block group (Active Comparator): The patients in external oblique intercostal plane block group will be received EOI plane block and patient controlled analgesia with morphine for postoperative analgesia
  Interventions: Other: Intravenous morphine patient control device; Other: External oblique intercostal plane block

INTERVENTIONS:
Other: Intravenous morphine patient control device — 24-hour morphine consumption will be recorded
Other: External oblique intercostal plane block — External oblique intercostal plane block will be administered before the surgery.
  Arms: External oblique intercostal plane block group

SUMMARY:
The external oblique intercostal (EOI) plane block is a novel approach upper abdominal wall analgesia. The EOI plane block can provide dermatomal sensory blockade of T6-T10 at the anterior axillary line and T6-T9 at the midline. It may be used for postoperative analgesia in obese patients because it is superficial and rapidly identifiable and performed in the supine position. the aim of this study is to investigate the postoperative analgesic efficacy of external oblique intercostal plane block in obese patients undergoing laparoscopic sleeve gastrectomy.

Researchers will compare the external oblique intercostal plane block group with control group to see if the EOI plane block is effective for postoperative analgesia in patients undergoing sleeve gastrectomy.

DETAILED DESCRIPTION:
Patients scheduled for elective laparoscopic sleeve gastrectomy will be separated into 2 groups: Control Group and External Oblique Intercostal Plane Block Group. Patients in Control Group will be received patient controlled analgesia with morphine for postoperative analgesia. Patients in External Oblique Intercostal Plane Block Group will be performed bilateral External Oblique Intercostal Plane Block before the surgery and received patient controlled analgesia with morphine for postoperative analgesia. Morphine consumption for first postoperative 24 hours, visual analog scale scores, time to need for first rescue analgesia, amount of rescue analgesic drug, incidence of postoperative nausea and vomiting will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* Patients with American Society of Anesthesiology (ASA) physical status II-III
* Patients scheduled for a laparoscopic sleeve gastrectomy

Exclusion Criteria:

* Allergy to local anesthetics
* Coagulopathy
* Skin infection at the EOI Plane Block area
* Advanced hepatic or renal failure
* Chronic pain syndromes
* Alcohol or drug abuse
* Severe pulmonary and/or cardiovascular disease
* Psychiatric disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-12-23 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | Postoperative 24 hours
  The amount of morphine required by the patient and given by the device will be recorded for the first 24 hours.

SECONDARY OUTCOMES:
Postoperative visual analog scale scores | Postoperative 24 hours
  Postoperative pain will be assessed using a visual analog scale (VAS) (from 0 = no pain to 10 = maximum possible pain) for the first 24 hours.
Time to first rescue analgesic | postoperative 24 hours
  The time for administration of first rescue analgesic will be recorded.
Rescue analgesic drug consumption | postoperative 24 hours
  The amount of rescue analgesic in mg required by the patient will be recorded for the first 24 hours.
Incidence of postoperative nausea and vomiting | postoperative 24 hours
  Number of patients developing postoperative nausea and vomiting will be recorded for the first 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ali Sait Kavakli, M.D., Principal Investigator — Istinye University; Taylan Sahin, M.D., Principal Investigator — Istinye University
Locations (1):
- Istinye University Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Kavakli AS, Sahin T, Koc U, Karaveli A. Ultrasound-Guided External Oblique Intercostal Plane Block for Postoperative Analgesia in Laparoscopic Sleeve Gastrectomy: A Prospective, Randomized, Controlled, Patient and Observer-Blinded Study. Obes Surg. 2024 May;34(5):1505-1512. doi: 10.1007/s11695-024-07174-9. Epub 2024 Mar 18. PMID 38499943